CLINICAL TRIAL: NCT01023646
Title: Evaluation of Glycemic Index to Assess Diet Associated Chronic Disease Risk
Brief Title: Glycemic Index - Variability Among Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: R01DK073321 (NIH); R01DK073321 (NIH)
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Diabetes; Obesity; Metabolic Syndrome; Cardiovascular Disease
Keywords: Glycemic Index; Glycemic Load; Glucose; Insulin; Lipoproteins; Free fatty acids
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Metabolic Syndrome; Cardiovascular Diseases; Insulin Resistance | interventions — Carbohydrates; Proteins; CD36 Antigens; Dietary Fiber

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- carbohydrate load (Other): Food challenge - Carbohydrate load
  Interventions: Other: Carbohydrate load
- Carbohydrate + Protein (Other): Food challenge - carbohydrate + protein
  Interventions: Other: Carbohydrate + Protein
- Carbohydrate + Fat (Other): Food challenge - carbohydrate + fat
  Interventions: Other: Carbohydrate + Fat
- Fiber (Other): Food challenge - carbohydrate + fiber
  Interventions: Other: Fiber

INTERVENTIONS:
Other: Carbohydrate + Protein — Light Tuna Packed in water.
  Arms: Carbohydrate + Protein
Other: Carbohydrate + Fat — Butter
  Arms: Carbohydrate + Fat
Other: Fiber — Unrefined Carbohydrate
  Arms: Fiber
Other: Carbohydrate load — Carbohydrate
  Arms: carbohydrate load

SUMMARY:
The purpose of this study is to determine the variability in glycemic index determinations for individual foods and food combinations. The study will also evaluate the changes in insulin and free fatty acid levels, plasma lipid and lipoprotein profiles, C-reactive protein-a marker of inflammation and glycosylated hemoglobin- a marker of glucose metabolism during a five-hour period after eating the food or foods. Additionally, supplementary data on variation in oral sensation, habitual food intake, food preferences and genes mediating sensory perception and dietary behaviors (supported by a grant from the Tufts Ross Aging Initiative) will be related to the outcomes on the present study.

DETAILED DESCRIPTION:
The objective of this proposal is to investigate the intra-individual reproducibility (within the same individual, when repeatedly measured) and inter-individual variability (among individuals) of glycemic index (GI) and glycemic load (GL) value determinations for individual foods and food combinations. The specific aims to accomplished this objective are to evaluate reproducibility and variability of GI value determinations in volunteers differing in biologic characteristics - body mass index (BMI), age and gender; assess the effect of macronutrient amounts and combinations, and fiber on variability of GI and GL value determinations; assess the effect of prior meal macronutrient composition ('second meal' effect) on GI value determinations; and relate these data to chronic disease risk factors monitored prior to and during the intervention period. These aims will be accomplished by assessing intra-individual reproducibility and inter-individual variability of repeated GI value determinations for white bread, commonly used as a reference food, relative to glucose, in volunteers selected to represent a range of BMI's (18-24.9, 25-29.9, 30-35) and ages (18-49.9, 50-85 y), and on the basis of gender, and relate these data to body composition and insulin sensitivity (Phase I). This work will then be extended to address issues related to variability potentially introduced by differences in macronutrient and fiber combinations and loads (Phase II), and finally by 'second meal' effects (Phase III). Prior to each set of food challenges (glucose and test food[s] in random order) volunteers will be characterized on the basis of fasting HbA1c; lipids and lipoproteins; insulin, glucose and C-reactive protein. During the 5-hour challenge (sampling at 0, 15, 30, 45, 60, and every 30 minutes thereafter) volunteers will be monitored for changes in blood glucose, insulin, triglycerides, total, low density lipoprotein and high density lipoprotein cholesterol, and non-esterified fatty acid levels. Additionally, supplementary data on variation in oral sensation, habitual food intake, food preferences and genes mediating sensory perception and dietary behaviors (supported by a grant from the Tufts Ross Aging Initiative) will be related to the outcomes on the present study. The concepts of both GI and GL are in the public domain and it has been suggested that the concepts be incorporated into U.S. federal dietary guidance (U.S. Dietary Guidelines and Dietary References Intakes) formulated to promote health and reduce chronic disease risk. This proposal addresses some of the understudied areas for which additional information would be useful in order to determine whether GI and GL should be used to classify foods on an individual basis, as has been suggested, and when formulating dietary guidance for the general population.

ELIGIBILITY:
Inclusion Criteria:

* For Phase 1 (Study 1) a total of seventy five volunteers will be included in the study. This study will be conducted in adult men and women (18-85 y) free of known chronic disease with BMI 18 to 35 kg/m2.
* For Phase 2 (Studies 2, 3, 4, and 5) a total of 80 volunteers will be included, 20 volunteers per study. Phase 2 studies will be conducted in adult men and women (50 - 85 y) free of known chronic disease and with a BMI of 25 to 35 kg/m2.
* For Phase 3 (Study 6) a total of 20 volunteers will be included in the study. Phase 3 study will be conducted in adult men and women (50-85 y) free of known chronic disease and with a BMI of 25 to 35 kg/m2.

Exclusion criteria:

* BMI ≥ 35 kg/m2 for Phase I, and BMI ≤ 25 to ≥ 35 kg/m2 for Phase II and III
* Renal disease, as defined by a history of chronic kidney disease or by glomerular filtration rate of < 60 ml.min/1.73 m2 calculated from screening blood tests.
* Liver disease, as defined by a history of chronic hepatitis B or C, cholestatic or cirrhotic liver disease, nonalcoholic fatty liver disease, elevations of serum glutamate pyruvate transaminase (SGPT) or serum glutamate oxaloacetate transaminase (SGOT) greater than 1.5 times the upper limit of normal at screening, bilirubin greater than 2 mg/dL (in the absence of benign causes of elevated bilirubin such as Gilbert's syndrome) at screening, or albumin below the lower limit of normal.
* Untreated hypertension, defined as systolic blood pressure (SBP) > 140 mm and diastolic blood pressure (DBP) > 90 mm.
* Irritable bowel syndrome.
* Malabsorptive disorder and inflammatory bowel disease.
* Disorders of esophageal and gastrointestinal motility, and previous esophageal or gastric resection.
* History of chronic pancreatitis, or history of acute pancreatitis within the last year.
* Hypothyroidism or hyperthyroidism, as defined as screening thyroid-stimulating hormone (TSH) outside of normal ranges.
* Anemia, as defined by screening hematocrit of 34% for women and 38% for men.
* Smoking within the past 6 months.
* Diabetes.
* Fasting glucose ≥ 125 mg/dL.
* Pregnancy.
* Breastfeeding.
* History of polycystic ovary syndrome
* History of autoimmune or other connective tissue disorders associated with chronic inflammation, such as rheumatoid arthritis.
* Alcohol consumption > 7 drinks/week.
* Use of medications or supplements known to affect glucose metabolism.
* Use of medications or supplements known to affect lipid metabolism.
* Established cardiovascular disease (myocardial infarction, stroke, heart failure, coronary artery. bypass graft, stenosis > 50%, peripheral arterial disease).
* Unwillingness to adhere to study protocol.
* Weight gain or loss of more than 15 lbs within 6 months prior to enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2007-12; Primary Completion 2015-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Glucose, Insulin, Free Fatty Acids. | 5 hours

SECONDARY OUTCOMES:
Fasting and non-fasting plasma lipids and lipoproteins, C reactive protein (CRP), HbAIc. | 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alice H Lichtenstein, D.Sc., Principal Investigator — JM USDA Human Nutrition Research Center on Aging at Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] Jenkins DJ, Wolever TM, Taylor RH, Barker H, Fielden H, Baldwin JM, Bowling AC, Newman HC, Jenkins AL, Goff DV. Glycemic index of foods: a physiological basis for carbohydrate exchange. Am J Clin Nutr. 1981 Mar;34(3):362-6. doi: 10.1093/ajcn/34.3.362. PMID 6259925
- [Background] Salmeron J, Manson JE, Stampfer MJ, Colditz GA, Wing AL, Willett WC. Dietary fiber, glycemic load, and risk of non-insulin-dependent diabetes mellitus in women. JAMA. 1997 Feb 12;277(6):472-7. doi: 10.1001/jama.1997.03540300040031. PMID 9020271
- [Background] Salmeron J, Ascherio A, Rimm EB, Colditz GA, Spiegelman D, Jenkins DJ, Stampfer MJ, Wing AL, Willett WC. Dietary fiber, glycemic load, and risk of NIDDM in men. Diabetes Care. 1997 Apr;20(4):545-50. doi: 10.2337/diacare.20.4.545. PMID 9096978
- [Background] Amano Y, Kawakubo K, Lee JS, Tang AC, Sugiyama M, Mori K. Correlation between dietary glycemic index and cardiovascular disease risk factors among Japanese women. Eur J Clin Nutr. 2004 Nov;58(11):1472-8. doi: 10.1038/sj.ejcn.1601992. PMID 15127092
- [Background] Schulze MB, Liu S, Rimm EB, Manson JE, Willett WC, Hu FB. Glycemic index, glycemic load, and dietary fiber intake and incidence of type 2 diabetes in younger and middle-aged women. Am J Clin Nutr. 2004 Aug;80(2):348-56. doi: 10.1093/ajcn/80.2.348. PMID 15277155
- [Background] Wolever TM, Csima A, Jenkins DJ, Wong GS, Josse RG. The glycemic index: variation between subjects and predictive difference. J Am Coll Nutr. 1989 Jun;8(3):235-47. doi: 10.1080/07315724.1989.10720298. PMID 2760355
- [Background] Wolever TM, Jenkins DJ, Josse RG, Wong GS, Lee R. The glycemic index: similarity of values derived in insulin-dependent and non-insulin-dependent diabetic patients. J Am Coll Nutr. 1987 Aug;6(4):295-305. doi: 10.1080/07315724.1987.10720191. PMID 3611527
- [Background] Jenkins DJ, Wolever TM, Wong GS, Kenshole A, Josse RG, Thompson LU, Lam KY. Glycemic responses to foods: possible differences between insulin-dependent and noninsulin-dependent diabetics. Am J Clin Nutr. 1984 Nov;40(5):971-81. doi: 10.1093/ajcn/40.5.971. PMID 6496392
- [Background] Foster-Powell K, Holt SH, Brand-Miller JC. International table of glycemic index and glycemic load values: 2002. Am J Clin Nutr. 2002 Jul;76(1):5-56. doi: 10.1093/ajcn/76.1.5. PMID 12081815
- [Background] Wolever TM, Vorster HH, Bjorck I, Brand-Miller J, Brighenti F, Mann JI, Ramdath DD, Granfeldt Y, Holt S, Perry TL, Venter C, Xiaomei Wu. Determination of the glycaemic index of foods: interlaboratory study. Eur J Clin Nutr. 2003 Mar;57(3):475-82. doi: 10.1038/sj.ejcn.1601551. PMID 12627186
- [Background] Wolever TM, Jenkins DJ. The use of the glycemic index in predicting the blood glucose response to mixed meals. Am J Clin Nutr. 1986 Jan;43(1):167-72. doi: 10.1093/ajcn/43.1.167. PMID 3942088
- [Background] Vega-Lopez S, Ausman LM, Griffith JL, Lichtenstein AH. Interindividual variability and intra-individual reproducibility of glycemic index values for commercial white bread. Diabetes Care. 2007 Jun;30(6):1412-7. doi: 10.2337/dc06-1598. Epub 2007 Mar 23. PMID 17384339
- [Derived] Meng H, Matthan NR, Ausman LM, Lichtenstein AH. Effect of prior meal macronutrient composition on postprandial glycemic responses and glycemic index and glycemic load value determinations. Am J Clin Nutr. 2017 Nov;106(5):1246-1256. doi: 10.3945/ajcn.117.162727. Epub 2017 Sep 13. PMID 28903959
- [Derived] Meng H, Matthan NR, Ausman LM, Lichtenstein AH. Effect of macronutrients and fiber on postprandial glycemic responses and meal glycemic index and glycemic load value determinations. Am J Clin Nutr. 2017 Apr;105(4):842-853. doi: 10.3945/ajcn.116.144162. Epub 2017 Feb 15. PMID 28202475
- [Derived] Matthan NR, Ausman LM, Meng H, Tighiouart H, Lichtenstein AH. Estimating the reliability of glycemic index values and potential sources of methodological and biological variability. Am J Clin Nutr. 2016 Oct;104(4):1004-1013. doi: 10.3945/ajcn.116.137208. Epub 2016 Sep 7. PMID 27604773